CLINICAL TRIAL: NCT04994717
Title: Phase 3 Randomized, Controlled Study of Blinatumomab Alternating With Low-intensity Chemotherapy Versus Standard of Care for Older Adults With Newly Diagnosed Philadelphia-negative B-cell Precursor Acute Lymphoblastic Leukemia With Safety Run-in (Golden Gate Study)
Brief Title: Study Comparing Blinatumomab Alternating With Low-intensity Chemotherapy Versus Standard of Care Chemotherapy for Older Adults With Newly Diagnosed Philadelphia-negative B-cell Precursor Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190360; 2023-503640-14 (EudraCT Number)
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Newly Diagnosed Philadelphia (Ph)-Negative B-cell Precursor Acute Lymphoblastic Leukemia (ALL)
Keywords: Newly Diagnosed Philadelphia (Ph)-negative B-cell Precursor Acute Lymphoblastic Leukemia (ALL); Blinatumomab; Low-intensity Chemotherapy; GMALL HyperCVAD
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-in: Blinatumomab alternating with low-intensity chemotherapy (Experimental): The safety run-in will be performed prior to initiating the phase 3 randomized part of the study. This safety run-in is to evaluate the safety and tolerability of blinatumomab alternating with low-intensity chemotherapy.
  The safety run-in also evaluates a shorter dose step interval from (4 days instead of 7 days) and a 1-week (instead of 2-week) drug free interval between blinatumomab cycles. Blinatumomab will be infused at a lower dose for 4 days and increase to a higher dose on Day 5 of the infusion for the remainder of the infusion.
  Interventions: Drug: Blinatumomab; Drug: Low-intensity chemotherapy regimen
- Phase 3: Blinatumomab alternating with low-intensity chemotherapy (Experimental): Participants will receive blinatumomab alternating with low-intensity chemotherapy.
  Interventions: Drug: Blinatumomab; Drug: Low-intensity chemotherapy regimen
- Phase 3: Standard of care (SOC) chemotherapy (Active Comparator): Participants will receive 1 of 2 SOC chemotherapy regimens (GMALL or HyperCVAD) per investigator's choice.
  Interventions: Drug: SOC chemotherapy regimen

INTERVENTIONS:
Drug: Blinatumomab — Continuous intravenous (cIV) infusion
  Other Names: Blincyto®
  Arms: Phase 3: Blinatumomab alternating with low-intensity chemotherapy; Safety Run-in: Blinatumomab alternating with low-intensity chemotherapy
Drug: Low-intensity chemotherapy regimen — Intravenous (IV), oral (PO), subcutaneous (SC), or intrathecal (IT) administration.
  Arms: Phase 3: Blinatumomab alternating with low-intensity chemotherapy; Safety Run-in: Blinatumomab alternating with low-intensity chemotherapy
Drug: SOC chemotherapy regimen — Intravenous (IV), oral (PO), subcutaneous (SC), or intrathecal (IT) administration.
  Arms: Phase 3: Standard of care (SOC) chemotherapy

SUMMARY:
The safety run-in part of the study aims to evaluate the safety and tolerability of blinatumomab alternating with low-intensity chemotherapy. The phase 3 part of the study aims to compare event-free survival (EFS) and overall survival (OS) of participants receiving blinatumomab alternating with low-intensity chemotherapy to EFS and (OS) of participants receiving standard of care (SOC) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 55 years at the time of informed consent. OR

Age 40 to < 55 years of age if at least 1 of the following comorbidities at the time of informed consent:

* history of grades 3 and 4 pancreatitis
* diabetes mellitus with end-organ damage
* severe liver disease such as cirrhosis stage 2 with portal hypertension or history of esophageal variceal bleeding and aspartate transaminase (AST)/alanine aminotransferase (ALT) > 10 x upper limit of normal (ULN) (liver cirrhosis must be confirmed by biopsy)
* body mass index (BMI) ≥ 40 combined with relevant comorbidities such as metabolic syndrome
* Any further combination of documented severe comorbidities that the investigator judges to be incompatible with administering an intensive pediatric based, adult adapted standard chemotherapy regimen but still compatible with the suggested protocol for older participants in both the experimental and the SOC arm. The participant history will be reviewed by the medical monitor during screening to determine enrollment acceptability based on a standard list with types of comorbidities allowed.

  * Participants with newly diagnosed Philadelphia (Ph)-negative B-cell precursor acute lymphoblastic leukemia (ALL)
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, higher ECOG score allowed if due to underlying leukemia
  * All participants must have adequate organ function as defined below:
* renal: estimated glomerular filtration rate based on MDRD calculation ≥ 50 mL/min/1.73 m^2
* liver function: total bilirubin ≤ 2x upper limit of normal (ULN; unless Gilbert's Disease or if liver involvement with leukemia); exception for participants 40 to < 55 years of age if they have a comorbidity listed above: severe liver disease such as cirrhosis stage 2 with portal hypertension or history of esophageal variceal bleeding and AST/ALT > 10 x ULN (liver cirrhosis must be confirmed by biopsy)
* cardiac: left ventricular ejection fraction (LVEF) ≥ 50% and no clinically significant, uncontrolled, or active cardiovascular disease (eg, myocardial infarction or stroke within 3 months). Consult with medical monitor as needed.

Exclusion Criteria:

* Active central nervous system (CNS) leukemia (i.e., CNS 3 leukemia, confirmed by lumbar puncture) not resolved with IT chemotherapy during screening.
* History of other malignancy within the past 3 years, with the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician Note: History of other malignancy (eg, multiple myeloma) treated with immunomodulatory drugs (eg, lenalidomide, thalidomide) in the past 3 years is an exclusion.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
* Clinically relevant CNS pathology or event such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychiatric conditions that preclude the use of high dose of corticosteroids
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Known infection with human immunodeficiency virus (HIV)
* Known infection with chronic or active infection with hepatitis B (eg, hepatitis b surface [HBs] antigen reactive or quantifiable hepatitis b virus [HBV] viral load) or hepatitis C virus (HCV) (eg, HCV RNA [qualitative] is detected).

Active hepatitis B and C based on the following results:

* positive for hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B)
* negative HepBsAg and positive for hepatitis B core antibody: negative HBV DNA by PCR result is necessary to enroll.
* positive Hepatitis C virus antibody (HepCAb): negative hepatitis C virus RNA by PCR result is necessary to enroll.

  * Participant with symptoms and/or clinical signs and/or radiographic and/or sonographic signs that indicate an acute or uncontrolled chronic infection.
  * Cancer chemotherapy for this newly diagnosed B cell ALL before the start of protocol-required therapy with the exception of IT chemotherapy or optional pre-phase (debulking) chemotherapy. Radiation to a spot lesion such as chloroma or lytic lesion of bone or vertebrae for pain or vertebral stabilization is allowed.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2029-09-07 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety run-in: Number of Participants who Experience Treatment-emergent Adverse Events (TEAEs) | Up to approximately 5 years
  Number and percentage of participants who experience one or more TEAE, serious TEAE, treatment-related adverse events, and adverse events of interest.
Phase 3: Event-free Survival (EFS) | Up to approximately 5 years
  Time from randomization (enrollment) until treatment failure, relapse or death from any cause, whichever is earlier.
  Treatment failure is defined as not achieving a hematological complete CR with MRD response <10-4 by the end of the initial disease assessment period.
  Relapse is defined as hematologic relapse, extramedullary relapse, and/or molecular relapse (MRD positivity >= 10^-3), whichever occurs earlier, in participants with prior achievement of hematologic CR with MRD response <10^-4.
  Participants without an event will be censored at their last evaluable disease assessment date.
Phase 3: Overall Survival (OS) | Up to approximately 5 years
  OS is defined as time from randomization (enrollment) until death due to any cause.

SECONDARY OUTCOMES:
Safety run-in: Complete Remission (CR) Rate by the End of Initial Disease Assessment Period | Baseline to Week 14
Safety run-in: Minimal Residual Disease (MRD) Response by the End of Initial Disease Assessment Period | Baseline to Week 14
  MRD response is defined as the percentage of participants who achieve a response of < 10^-4 measured by polymerase chain reaction (PCR).
Safety run-in: Relapse-free Survival (RFS) | Up to approximately 5 years
  RFS: In participants who achieve CR, the time from first achievement of this response until date of the first relapse including hematologic relapse, extramedullary relapse, or death due to any cause, whichever occurs first.
Safety run-in: Minimal Residual Disease (MRD) Relapse Free Survival (RFS) | Up to approximately 5 years
  MRD RFS: In participants who achieve CR with MRD response, the time from first achievement of this response until date of of the first relapse including molecular relapse, hematological relapse, and/or extramedullary relapse, or death due to any cause, whichever occurs first. (Molecular relapse will be defined 2 ways: MRD>= 10^-3 and MRD>=10^-4. Participants without an event will be censored at their last evaluable disease assessment date.
Safety run-in: Steady State Concentration (Css) of Blinatumomab | Up to approximately 34 weeks
Safety run-in: Clearance (CL) of Blinatumomab | Up to approximately 34 weeks
Phase 3: Change from Baseline to End of Initial Disease Assessment Period in Fatigue Score | Baseline to Week 14
  Fatigue score will be measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - Short Form 7a.
Phase 3: Change from Baseline to End of Initial Disease Assessment Period in Pain Score | Baseline to Week 14
  Pain score will be measured by Brief Pain Inventory - Short Form (BPI-SF); Item 3: pain at its worst in the last 24 hours.
Phase 3: Change from Baseline to End of Initial Disease Assessment Period in Global Health Status | Baseline to Week 14
  Global health status will be measured by the Quality of Life Questionnaire (QLQ)-C30 global health status quality of life scale.
Phase 3: Change from Baseline to End of Initial Disease Assessment Period in Physical Function | Baseline to Week 14
  Physical function will be measured by the QLQ-C30 functional scale.
Phase 3: Change from Baseline to End of Initial Disease Assessment Period in Nausea and Vomiting | Baseline to Week 14
  Nausea and vomiting will be measured by the QLQ-C30 symptom scale.
Phase 3: Complete Remission (CR) Rate by the End of Initial Disease Assessment Period | Baseline to Week 14
Phase 3: Minimal Residual Disease (MRD) Response by the End of Initial Disease Assessment Period | Baseline to Week 14
  MRD response is defined as the percentage of participants who achieve a response of < 10^4 measured by polymerase chain reaction (PCR).
Phase 3: Relapse-free Survival (RFS) | Up to approximately 5 years
  RFS: In participants who achieve CR, the time from first achievement of this response until the date of the first relapse including hematologic relapse, extra medullary relapse, or death due to any cause, whichever occurs first. Participants without an event will be censored at their last evaluable disease assessment date.
Phase 3: Minimal Residual Disease (MRD) Relapse Free Survival (RFS) | Up to approximately 5 years
  In participants who achieve CR with MRD response, the time from first achievement of this response until date of the first relapse including molecular relapse, hematologic relapse, and/or extramedullary relapse, or death due to any cause, whichever occurs first. Molecular relapse will be defined 2 ways: MRD>= 10^-3 and MRD>= 10^-4. Participants without an event will be censored at their last evaluable disease assessment date
Phase 3: Minimal Residual Disease (MRD) Over Time | Up to approximately 5 years
Phase 3: Number of Participants who Experience Treatment-emergent Adverse Events (TEAEs) | Up to approximately 5 years
  Number and percentage of participants who experience one or more TEAE, serious TEAE, treatment-related adverse events, and adverse events of interest.
Phase 3: Number of Participants who Experience Cluster of Differentiation (CD) 19 Positive and Negative Relapse by Flow Cytometry for Bone Marrow | Up to approximately 5 years
Phase 3: Number of Participants who Experience Cluster of Differentiation (CD) 19 Positive and Negative Relapse Identified by Immunohistochemistry or Flow Cytometry for Cerebrospinal Fluid | Up to end of safety follow up (approximately 44 months)
Phase 3: Number of Participants who Experience Cluster of Differentiation (CD) 19 Positive and Negative Relapse for Extramedullary Sites other than Cerebrospinal Fluid | Up to end of safety follow up (approximately 44 months)
Phase 3: Rate of Lineage Switch to Acute Myeloid Leukemia (AML) | Up to end of safety follow up (approximately 44 months)
Phase 3: Localization of Relapse by Clinical Assessment | Up to end of safety follow up (approximately 44 months)
Phase 3: Mortality Rate in Participants who Experience Complete Remission (CR) | Up to approximately 5 years
Phase 3: Number of Participants who have Allogeneic Hematopoietic Stem Cell Transplant (alloHSCT) in Participants who Experience Continuous First Complete Remission (CR) | Up to approximately 5 years
Phase 3: Mortality Rate in Participants who Experience Complete Remission (CR) after Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT) | Up to approximately 5 years
Phase 3: Relapse Rate Following Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT) | Up to approximately 5 years
Phase 3: Time to Deterioration using the Fatigue Score | Up to approximately 5 years
  Fatigue score will be measured by PROMIS Fatigue-Short Form 7a.
Phase 3: Time to Improvements using the Fatigue Score | Up to approximately 5 years
  Fatigue score will be measured by PROMIS Fatigue-Short Form 7a.
Phase 3: Time to Deterioration using the Pain Score | Up to approximately 5 years
  Pain score will be measured by BPI-SF; Item 3: pain at its worst in the last 24 hours.
Phase 3: Time to Improvements using the Pain Score | Up to approximately 5 years
  Pain score will be measured by BPI-SF; Item 3: pain at its worst in the last 24 hours.
Phase 3: Change from Baseline in Global Health Status, Physical Function, Nausea/Vomiting, and All Other Subscales of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline to end of study (up to approximately 5 years)
  EORTC QLQ-C30 will include global health status, physical functioning, emotional functioning, cognitive functioning, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, diarrhea, and financial difficulties will be measured by EORTC QLQ-C30.
Phase 3: Time to Deterioration for Global Health Status, Physical Function, Nausea/Vomiting, and All Other Subscales of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Up to approximately 5 years
  Global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, diarrhea, and financial difficulties will be measured by EORTC QCQ-C30.
Phase 3: Time to Improvements for Global Health Status, Physical Function, Nausea/Vomiting, and All Other Subscales of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Up to approximately 5 years
  Global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, diarrhea, and financial difficulties will be measured by EORTC QCQ-C30.
Steady State Concentration of Blinatumomab | Up to approximately Day 36
Clearance of Blinatumomab | Up to approximately Day 36

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (192):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of California Irvine, Orange, California
  - University of California San Francisco, San Francisco, California
  - Adventist Health System/Sunbelt, Inc d/b/a AdventHealth Orlando, Orlando, Florida
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Saint Francis Hospital, Inc, Greenville, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (13):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (4):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Ordensklinikum Linz Elisabethinen, Linz
  - Hanusch Krankenhaus, Vienna
- Belgium (9):
  - Institut Jules Bordet, Anderlecht
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - AZ Delta Campus Rumbeke, Roeselare
  - Centre Hospitalier Universitaire-Universite Catholique de Louvain Namur-Site Godinne, Yvoir
- Brazil (8):
  - Igesd Instituto de Gestao Estrategica da Saude do Distrito Federal, Brasília, Federal District
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundacao Amaral Carvalho, Jaú, São Paulo
  - Hosp Clin Fac Med Ribeirao Preto Usp, Ribeirão Preto, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São Jose Do Rio Preto, São Paulo
  - Hemorio, Rio de Janeiro
  - Instituto Cancer Sao Paulo Icesp, São Paulo
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Specialized Hospital for Active Treatment of Hematology Diseases EAD, Sofia
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II, Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CEMTL Hopital Maisonneuve Rosemont, Montreal, Quebec
- Chile (3):
  - Fundacion Arturo Lopez Perez, Santiago
  - Inmunocel, Santiago
  - Clinica Alemana de Santiago, Santiago
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Ustav hematologie a krevni transfuze, Prague
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Odense
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- France (14):
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Dijon - Hopital du Bocage, Dijon
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, Le Chesnay
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire de Nantes - Hopital Hotel Dieu, Nantes
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Hopital Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - Universitaetsklinikum Augsburg, Augsburg
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein - Kiel, Kiel
  - Klinikum der LMU Muenchen, München
- Greece (8):
  - Evangelismos Hospital, Athens
  - Laiko General Hospital of Athens, Athens
  - Attiko General University Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - General Hospital of Thessaloniki Georgios Papanikolaou, Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Princess Margaret Hospital, Kowloon
  - Tuen Mun Hospital, New Territories
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Heves Varmegyei Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
- Israel (3):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
- Italy (13):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni xxiii, Bergamo
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola, Bologna
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Azienda Unita Sanitaria Locale LE Presidio Ospedaliero Vito Fazzi Polo Oncologico Giovanni Paolo II, Lecce
  - Azienda Unità Locale Socio Sanitaria 3 Ospedale Dell Angelo, Mestre (VE)
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Unita Sanitaria Locale Pescara Ospedale Civile Santo Spirito, Pescara
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Azienda Ospedaliero Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata di Verona Ospedale G B Rossi Borgo Roma, Verona
- Japan (23):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Tesshokai Kameda General Hospital, Kamogawa-shi, Chiba
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gunma Saiseikai Maebashi Hospital, Maebashi, Gunma
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Kindai University Hospital, Sakai-shi, Osaka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
- Mexico (5):
  - Boca Clinical Trials Mexico SC, Mexico City, Mexico City
  - Centro Oncologico Internacional, Mexico City, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Hematologica Alta Especialidad, Huixquilucan
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Portugal (5):
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Unidade Local de Saude de Sao Jose, EPE - Hospital de Santo Antonio dos Capuchos, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (6):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica sv Cyrila a Metoda, Bratislava
- South Korea (7):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (9):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complejo Asistencial Universitario de Salamanca Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Institut Catala d Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario 12 de Octubre, Madrid
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Inselspital Bern, Bern, Switzerland
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Turkey (Türkiye) (6):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Memorial Antalya Hastanesi, Antalya
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (2):
  - University College London, London
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com